CLINICAL TRIAL: NCT06833476
Title: Transcatheter Tricuspid Valve Replacement (TTVR) in Patients With Severe TR ONgoing Evidence Generation (STRONG) Under Coverage With Evidence Development (CED)
Brief Title: TTVR STRONG Under Coverage With Evidence Development (CED) Study
Acronym: STRONG
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: EVOQUE CED
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation
Keywords: EVOQUE; Coverage with Evidence Development; CED; TVT Registry
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- EVOQUE treated: Medicare patients with at least severe Tricuspid Regurgitation who received a Transcatheter Tricuspid Valve Replacement with the EVOQUE device and is identified in the TVT Registry
  Interventions: Other: EVOQUE
- EVOQUE eligible: Medicare eligible patients with severe, symptomatic Tricuspid Regurgitation that are identifiable in a commercial claims database linked with electronic health records.

INTERVENTIONS:
Other: EVOQUE — This is a retrospective, non-randomized study. The decision to intervene by TTVR with the EVOQUE device is made by the heart team.
  Groups: EVOQUE treated

SUMMARY:
This Coverage with Evidence Development (CED) study measures the long-term health outcomes of patients with severe, symptomatic Tricuspid Regurgitation who received a Transcatheter Tricuspid Valve Replacement procedure using the EVOQUE system.

DETAILED DESCRIPTION:
This is a retrospective, non-randomized cohort study measuring 2-year effectiveness of the EVOQUE Transcatheter Tricuspid Valve Replacement (TTVR) system in the real-world.

This study will retrospectively evaluate EVOQUE treated patients in the STS/ACC TVT Registry who have at least severe Tricuspid Regurgitation and can be deterministically linked with Medicare data.

This group will be compared to Medicare eligible and EVOQUE eligible patients evaluated in a standard of care setting from a commercial claims database linked with electronic health records.

We will evaluate the primary outcome measure in various subgroups.

There will be continued access enrollment after the primary completion date.

ELIGIBILITY:
Inclusion Criteria:

Medicare eligible patients who have received an EVOQUE device or are EVOQUE eligible and have at least severe Tricuspid Regurgitation

Exclusion Criteria:

Commercially insured patients who have received an EVOQUE device or are EVOQUE eligible or Medicare eligible patients with less than severe Tricuspid Regurgitation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Medicare eligible real-world patients with severe, symptomatic tricuspid regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 2044 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite (All-Cause Death or Heart Failure Hospitalization) | 2 years
  Time to death or heart failure hospitalization after time zero

CONTACTS AND LOCATIONS:
Locations (1):
- Edwards Lifesciences, Irvine, California, United States